CLINICAL TRIAL: NCT03723668
Title: Kidney Transplant Outcome and Organ Acceptance Practice Pattern: A Nationwide Analyses in the US and France
Acronym: USFRKT
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: University of Pennsylvania (Other); Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Other Study IDs: USFRKT1
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Kidney Failure; Transplant;Failure,Kidney
Keywords: kidney transplantation; allograft survival
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OPTN data system: In the US, data on the donors and kidney transplant recipients will be obtained using registry data from the Organ Procurement and Transplantation Network (OPTN). The OPTN data system includes data on all donors, waitlisted candidates, and transplant recipients in the US, as submitted by the members of the Organ Procurement and Transplantation Network. The Health Resources and Services Administration (HRSA) of the US Department of Health and Human Services oversees the activities of the OPTN contractor.
- CRISTAL registry: In France, data on the donors and recipients in the French cohort will be obtained from the national CRISTAL registry, initiated in 1996 and maintained by the Agence de la Biomédecine, which prospectively collects data on all potential donors and organ transplant candidates, along with their outcomes. By law, data collection is provided by all organ procurement organizations and transplant centers in France; research studies based on the national CRISTAL registry are part of the transplant assessment activities and do not require institutional review board approval.

SUMMARY:
Despite the considerable advances in short-term outcomes, kidney transplant recipients continue to suffer from late allograft failure, and little improvement has been made over the past 15 years. The worldwide scarcity of donated kidneys and the decline in the number of living donor transplants have prompted a variety of efforts to expand the organ supply, such as accepting organs from donors who were older or had comorbidities or other injuries.

Two major initiatives from the United Network for Organ Sharing (UNOS), the organization responsible for organ allocation in the US, failed to improve the kidney acceptance rate. First, UNOS introduced the Kidney Donor Risk Index (KDRI) for all kidney offers in 2012. The KDRI is a score that predicts survival of deceased donor kidneys based on 10 donor characteristics and was intended to simplify the process of judging organ quality for clinicians. Second, in 2014, UNOS changed the kidney allocation system so that lower-quality kidneys are offered over wider geographic areas. Despite the ongoing severe organ shortage and these allocation initiatives, the number of discarded kidneys rose from 2,127 (14.9%) in 2006 to 3,631 (20%) in 2016. In this context, the experience of transplant programs outside the US could offer novel approaches to making organ utilization more efficient through the examination of the disposition of organs that are usually discarded in the US.

This project aims:

1. To evaluate the potential benefit of transplanting kidneys that would have been discarded otherwise in the US
2. Computer simulation models on real life data to estimate the number of kidney transplants that would have taken place using data from a nationwide cohort study in two countries (France, the US);
3. To evaluate the potential gains in allograft survival years that would result in the US from a less restrictive kidney acceptance practice such as the one from France.

DETAILED DESCRIPTION:
Background The worldwide scarcity of donated kidneys and the decline in the number of living donor transplants have prompted a variety of efforts to expand the organ supply, such as accepting organs from donors who were older or had comorbidities or other injuries. This study aims to simulate the application of allocation policies from the US to France and vice-versa in two comprehensive cohorts.

Main Outcome(s) and Measure(s)

In the US, data on the donors and kidney transplant recipients will be obtained using registry data from the Organ Procurement and Transplantation Network (OPTN). The OPTN data system includes data on all donors, waitlisted candidates, and transplant recipients in the US, as submitted by the members of the Organ Procurement and Transplantation Network. The Health Resources and Services Administration (HRSA) of the US Department of Health and Human Services oversees the activities of the OPTN contractor.

In France, data on the donors and recipients in the French cohort will be obtained from the national CRISTAL registry, initiated in 1996 and maintained by the Agence de la Biomédecine, which prospectively collects data on all potential donors and organ transplant candidates, along with their outcomes. By law, data collection is provided by all organ procurement organizations and transplant centers in France; research studies based on the national CRISTAL registry are part of the transplant assessment activities and do not require institutional review board approval.

Graft survival will be estimated using the Kaplan-Meier method. Duration of follow-up started with the patient risk evaluation (starting point) up to the date of the kidney graft loss, defined as a patient's return to dialysis, or retransplantation. For patients who died with a functioning graft, graft survival will be censored at the time of death.

The investigators will then model kidney allograft discard practices using KDRI and perform simulation to estimate kidneys that would have been discarded in each country using the discard score (Monte-Carlo technique). The investigators will also quantify predicted kidney allograft survival of the discarded kidneys. Eventually, the investigators will estimate the gain of allograft life years based on observed survival data.

Groups/Cohorts

All kidney transplantation occurring in France and in the US from 2004 to 2014 with available data to calculate the KDRI and the Kidney Donor Profile Index (KDPI), with lower values suggestive of better quality. The KDRI and KDPI are currently used as part of the OPTN allocation system for deceased donor kidneys in the US and have been validated as reliable measures of organ quality in the US.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive kidneys recovered for the purpose of transplantation from donors deceased from brain death or circulatory death,
* Between January 1, 2004 and December 31, 2014.

Exclusion Criteria:

* Living renal transplants,
* Multiorgan transplant recipients,
* Kidneys offered to transplant centers but never recovered, and
* Patients with missing data to calculate the KDRI score

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All kidney transplantation occurring in France and in the US from 2004 to 2014 with available data to calculate the KDRI and the Kidney Donor Profile Index (KDPI), with lower values suggestive of better quality. The KDRI and KDPI are currently used as part of the OPTN allocation system for deceased donor kidneys in the US and have been validated as reliable measures of organ quality in the US.
Sampling Method: Probability Sample
Enrollment: 94017 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Number of kidneys procured and discarded. | 10 years
  In some instances, the two kidneys might be procured from one donor but one or both kidneys may eventually be discarded and thus, not transplanted. This information was retrieved in both the OPTN data system and CRISTAL registry.

SECONDARY OUTCOMES:
Probability of allograft failure after transplantation. | 10 years
  This is defined as the need for renal replacement therapy or preemptive re-transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reese, MD, Principal Investigator — Kidney Transplantation Care at Veteran's Affairs Medical Center; Alex Loupy, Principal Investigator — Paris Transplant Group, INSERM, UMR-S970, Paris, France
Locations (2):
- Kidney Transplantation Care at Veteran's Affairs Medical Center, Philadelphia, Pennsylvania, United States
- Paris Transplant Group, Paris, France

REFERENCES:
- [Derived] Aubert O, Reese PP, Audry B, Bouatou Y, Raynaud M, Viglietti D, Legendre C, Glotz D, Empana JP, Jouven X, Lefaucheur C, Jacquelinet C, Loupy A. Disparities in Acceptance of Deceased Donor Kidneys Between the United States and France and Estimated Effects of Increased US Acceptance. JAMA Intern Med. 2019 Oct 1;179(10):1365-1374. doi: 10.1001/jamainternmed.2019.2322. PMID 31449299